CLINICAL TRIAL: NCT05312229
Title: Implementing and Sustaining Critical Time Intervention (CTI) in Case Management Programs for Homeless-experienced Veterans (PII 21-285)
Brief Title: Housing Transitions QUERI
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, Los Angeles (Other); Center for the Advancement of Critical Time Intervention (Unknown); University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PIX 22-001; PII 21-285 (Other Grant/Funding Number: QUERI)
Record Dates: First submitted 2022-03-10; First posted 2022-04-05 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Homelessness
Keywords: Care Management; Homeless; Implementation; Mental Health Care; Quality Assurance, Improvement

STUDY DESIGN:
Intervention Model Description: The investigators are implementing Critical Time Intervention (CTI), an evidence-based, time limited case management practice for individuals experiencing homelessness. The investigators will be randomizing sites receiving CTI into one of two levels of implementation support (low vs. high intensity support).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Replicating Effective Programs (REP) (Experimental): A stakeholder-informed training and technical assistance implementation strategy
  Interventions: Behavioral: Critical Time Intervention; Other: Replicating Effective Programs
- REP + External Facilitation (Enhanced REP) (Active Comparator): REP plus site specific weekly facilitation to support CTI implementation.
  Interventions: Behavioral: Critical Time Intervention; Other: External Facilitation; Other: Replicating Effective Programs
- Control Group (No Intervention): No CTI implementation

INTERVENTIONS:
Behavioral: Critical Time Intervention — An evidence-based, structured, and time-limited case management practice
  Other Names: CTI
  Arms: REP + External Facilitation (Enhanced REP); Replicating Effective Programs (REP)
Other: External Facilitation — Site-specific support to help sites develop tailored plans to implement CTI.
  Other Names: Coaching
  Arms: REP + External Facilitation (Enhanced REP)
Other: Replicating Effective Programs — A stakeholder-informed training and technical assistance implementation strategy
  Other Names: REP
  Arms: REP + External Facilitation (Enhanced REP); Replicating Effective Programs (REP)

SUMMARY:
The VA Grant and Per Diem (GPD) case management aftercare program provides six months of case management for homeless-experienced Veterans undergoing housing transitions. This Partnered Implementation Initiative (PII) proposes to implement and evaluate Critical Time Intervention (CTI)-an evidence-based, structured, and time-limited case management practice-in 32 GPD case management aftercare sites across the nation.

DETAILED DESCRIPTION:
The VA Grant and Per Diem case management (GPD-CM) program provides six months of case management for homeless-experienced Veterans (HEVs) undergoing housing transitions. At present, no specific case management paradigm is required in the GPD-CM program, resulting in practice variation across sites. This Partnered Implementation Initiative (PII) implements Critical Time Intervention (CTI)-an evidence-based, structured, and time-limited case management practice-at 32 VA GPD-CM sites. The investigators will use the Replicating Effective Programs (REP) implementation bundle to support CTI implementation at all 32 sites. Half of these sites will also receive 9 months of external facilitation (enhanced REP) as additional support for CTI implementation. In a type 3 hybrid trial, the investigators will use mixed methods to examine the impacts of REP versus enhanced REP. Using trial data, the investigators will develop a business case analysis and implementation playbook for the investigators' program partners to support continued CTI spread and sustainment in the GPD-CM program.

ELIGIBILITY:
Inclusion Criteria:

* Grant and Per Diem (GPD) case management aftercare grantees in 7 Veterans Integrated Service Networks (VISN), all of whom provide 6-months of case management to Veterans who have experienced homelessness.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Fidelity to CTI | 12 months after implementation start
  % of Sites with adequate fidelity to CTI at 12 months, as measured by the CTI fidelity scale
Sustainment of CTI | 18 months after implementation start
  % of Sites with adequate fidelity to CTI at 18 months, as measured by the CTI fidelity scale
Dollars spent delivering CTI at each site | Between 6 and 18 months after implementation start
  Case manager salary and benefits

SECONDARY OUTCOMES:
Housing stability | Between 6 and 18 months after implementation start
  Days between entry into the GPD case management program and indicator of housing instability
Cost of CTI as Implemented | Between 6 and 18 months after implementation start
  Mean monthly cost of CTI case management per GPD case management Veteran served, compared to the mean monthly cost in the non-CTI GPD case management programs.
Hospitalization rates | Between 6 and 18 months after implementation start
  Number of days between entry into the GPD case management program and hospitalization, number of hospitalizations, number of bed days
Cost of Implementation Strategies | Through study completion, 4 years
  Dollars spent on REP versus enhanced REP
Return on Investment (ROI) of CTI | 6-, 12-, and 18-months after GPD case management program enrollment
  Dollars saved via improved housing stability and decreased hospitalizations among patients engaged in CTI versus control participants
Outpatient service use | Between 6 and 18 months after implementation start
  Number of outpatient appointments

CONTACTS AND LOCATIONS:
Overall Officials: Sonya Emi Gabrielian, MD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Gabrielian S, Finley EP, Ganz DA, Barnard JM, Jackson NJ, Montgomery AE, Nelson RE, Cordasco KM. Comparing two implementation strategies for implementing and sustaining a case management practice serving homeless-experienced veterans: a protocol for a type 3 hybrid cluster-randomized trial. Implement Sci. 2022 Oct 3;17(1):67. doi: 10.1186/s13012-022-01236-1. PMID 36192785
- See also: Resources for VA Grant and Per Diem (GPD) case management aftercare grantee sites to implement and sustain Critical Time Intervention (CTI) at their sites. — https://www.VACTItoolkit.com